CLINICAL TRIAL: NCT06553677
Title: Clinical Evaluation of Tunneled Coronally Advanced Flap (TCAF) Versus Coronally Advanced Flap (CAF) Combined With Connective Tissue Graft in the Treatment of Isolated RT2 Gingival Recession Sites: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Tunneled Coronally Advanced Flap v.s Coronally Advanced Flap With Graft for Gingival Recession
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Hazem Mohamed Said Sallam, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Perio2804
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Gingival Recession, Localized
Keywords: TCAF; CAF; RT2; Gingival recession depth reduction
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: It's randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tunneled coronal advanced flap with connective tissue graft (Experimental): TCAF involves the elevation of one trapezoidal surgical papilla at the papilla with less interproximal clinical attachment loss, by a slightly divergent vertical incision extending beyond the mucogingival junction is done then a horizontal incision at a distance equal to the recession depth plus 1 mm apical to the papilla tip just as the conventional coronally advanced flap (CAF). Then a tunneling knife will be used to perform the intra-sulcular incision on the treated site and on the tooth adjacent to the papilla that will be preserved for tension-free flap advancement.
  The midfacial aspect of the tooth will be elevated with tunneling knives while the surgical papilla will be elevated in a split-thickness manner.
  . The anatomical papilla will be de-epithelialized, either with a surgical blade or micro scissors, while the other papilla will be gently mobilized with a tunneling instrument. .
  The harvested connective tissue graft will be inserted underneath the flap
  Interventions: Procedure: Tunneled coronal advanced flap with connective tissue graft
- Coronally advanced flap with connective tissue graft (Active Comparator): A trapezoidal-shaped flap will be elevated with a split-full-split approach in the coronal-apical direction:
  * The surgical papillae will be elevated by split thickness keeping the blade almost parallel to the root.
  * The soft tissue apical to the root exposure will be elevated in a full thickness manner to expose 3-4mm of bone apical to the bone dehiscence. This was done to include the periosteum in the thickness of that central portion of the flap covering the avascular root exposure.
  * The releasing vertical incisions will be elevated by split thickness keeping the blade parallel to the bone thus leaving the periosteum to protect the underlying bone in the lateral areas of the flap.
  * The part of the flap apical to bone exposure will be elevated by split-thickness, this step will be done so it is possible to move the flap passively in the coronal direction.
  The harvested connective tissue graft will be inserted underneath the flap
  Interventions: Procedure: Coronally advanced flap with connective tissue graft

INTERVENTIONS:
Procedure: Tunneled coronal advanced flap with connective tissue graft — Tunneled coronal advanced flap with connective tissue graft to treat isolated RT2 gingival recession sites.
  Arms: Tunneled coronal advanced flap with connective tissue graft
Procedure: Coronally advanced flap with connective tissue graft — Coronally advanced flap with connective tissue graft to treat isolated RT2 gingival recession sites
  Arms: Coronally advanced flap with connective tissue graft

SUMMARY:
The goal of this clinical trial is to evaluate gingival recession depth reduction using tunneled coronally advanced flap compared to coronally advanced flap, both combined with connective tissue graft in patients with isolated RT2 gingival recession sites.

DETAILED DESCRIPTION:
Gingival recession can cause clinical conditions that could be of main concern for patients. Techniques aiming for coverage of the gingival recession aim to address dentin hypersensitivity, non-carious cervical lesions (NCCLs) and enhance patient's esthetics (Cortellini & Bissada, 2018). Mid-buccal gingival recessions have been associated with patient's esthetic discomfort (Zucchelli & Mounssif, 2015). Most of the studies in the literature focus on the treatment of RT1 recession as they have the most favorable prognosis of full root coverage (Barootchi et al., 2020). Despite most studies focusing their attention on RT1 cases, RT2 defects are found to be the most prevalent type with 88.8% among patients according to (Romandini et al., 2020).

The coronally advanced flap and the tunneling technique are the most commonly performed surgical approaches for treating gingival recessions. However, these two approaches have commonly been regarded as alternatives to each other, with clinicians choosing to perform only one of them during root coverage procedures.

(Barootchi & Tavelli, 2022) aimed in his conducted case series to designate a surgical technique to treat isolated RT2 gingival recession defects in which he was trying to achieve and combine the advantage of both better access and graft stabilization in CAF and the preservation of the integrity of the papilla and better blood supply to the graft present in tunneling technique. The study concluded that the combination of both techniques in the same surgical design can have the potential to enhance flap and graft vascularization and improve clinical, esthetic, and patient-reported outcomes. To our knowledge, there is no conducted randomized clinical trials comparing the tunneled coronally advanced flap technique to the coronally advanced flap for gingival depth reduction.

So, this clinical trial aims to address this gap of the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 years or older.
2. Isolated recession defect classified as RT2.
3. Patients with healthy systemic condition.
4. Clinical indication and/or patient request for root coverage.
5. O'Leary index less than 20%.

Exclusion Criteria:

1. Pregnant females
2. Smokers: a contraindication for any plastic periodontal surgery.
3. Unmotivated and uncooperative patients with poor oral hygiene
4. Patients with habits that may compromise the longevity and affect the result of the study as alcoholism or parafunctional habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Gingival Recession Depth | 6 months
  It's measured as the distance between cemento-enamel junction (CEJ), and gingival margin (GM) using periodontal probe.

SECONDARY OUTCOMES:
Percentage of mean root coverage (MRC%) | 6 months
  (Preoperative vertical recession depth - Postoperative vertical recession/preoperative vertical recession) x 100 [%]
Percentage of complete root coverage (CRC%) | 6 months
  Number of defect sites with complete root coverage/ Total number of recession sites treated x 100 [%]
Gingival Recession Width | 6 months
  Measured at the widest point (it is the distance between the mesial gingival margin and the distal gingival margin of the tooth)
Gingival Thickness | 6 months
  Measured using transgingival needle probing using anesthesic needle a rubber stopper
Keratinized Tissue Width | 6 months
  Measured as the distance between the gingival margin and the mucogingival junction (MGJ).
Clinical Attachment Level | 6 months
  Measured from the CEJ to the bottom of the gingival sulcus.
Probing Pocket Depth | 6 months
  Measured from the gingival margin to the bottom of the gingival sulcus.
Pink Esthetic Score | 6 months
  It's a score by (Fürhauser et al., 2005) based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture.
  Each variable is assessed with a 0-1-2 score, with 2 being the best and 0 being the poorest score.
Post-operative pain | 2 weeks
  Visual Analogue Scale (VAS) with numerical scale from 0 to 10 ('no pain' to 'worst pain imaginable') measured daily for the first 2 weeks postoperatively.
Post-operative patient satisfaction | 2 weeks, 6 months
  A 3-item questionnaire will be given to the patients to be answered using a 7-point answer scale for assessing their satisfaction with the whole surgical procedure and the achieved results of the procedure performed.
Root coverage esthetic score | 6 months
  (Cairo et al., 2009) This score evaluates five variables: level of the gingival margin (GM) , marginal tissue contour (MTC), soft tissue texture (STT) , mucogingival junction (MGJ) alignment , and gingival color (GC).
  * GM: Zero point for failure of root coverage (gingival margin apical or equal to the baseline recession); 3 points partial root coverage; 6 points CRC.
  * MTC: Zero point irregular gingival margin (does not follow the CEJ); 1 point -proper marginal contour/ scalloped gingival margin (follows the CEJ).
  * STT: Zero point for scar formation and/or keloid-like appearance; I point absence of scar or keloid formation.
  * MGJ: Zero point -MGJ not aligned with the MGJ of adjacent teeth; 1 point if the MGJ aligned with the MGJ of adjacent teeth.
  * GC: Zero point color of tissue varies from gingival color at adjacent teeth; 1 point normal color and integration with the adjacent soft tissues.
    10 is the ideal esthetic score

CONTACTS AND LOCATIONS:
Overall Officials: Engy Ahmed, PhD, Study Chair — Cairo University; Omar A Ashour, PhD, Study Chair — Cairo University; Yehia H Amer, PhD, Study Chair — Cairo University; Omar H Sallam, MSc, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
I will check with my study chair.

REFERENCES:
- [Result] Barootchi S, Tavelli L. Tunneled coronally advanced flap for the treatment of isolated gingival recessions with deficient papilla. Int J Esthet Dent. 2022 Feb 17;17(1):14-26. PMID 35175005